CLINICAL TRIAL: NCT00291772
Title: Continuous Subcutaneous Infusion of Pramlintide and Insulin: A Randomized, Crossover Design Study
Brief Title: Continuous Subcutaneous Infusion of Pramlintide and Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sponsored Programs, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-17339
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; hypoglycemia; hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia | interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pramlintide — Basal and bolus pramlintide subcutaneous infusion
  Other Names: Symlin

SUMMARY:
The purpose of this study is to see if giving the study drug in a slow and steady dose will lower blood sugars during the meal and after-meal time.

DETAILED DESCRIPTION:
The Diabetes Control and Complications Trial (DCCT) showed that improving blood sugar control for individuals with Type 1 diabetes (T1DM) stopped or delayed the onset of long-term health problems. Insulin management is aimed to control blood sugar as near to normal as safely possible. However, the possibility of low blood sugars still remains. Low blood sugars the major limiting factor in gaining "tight" control of blood sugar. Insulin (the hormone that lowers blood sugar) and glucagon (hormone that raises blood sugar) play a key role in keeping this careful balance. There is a lack of insulin and failure of glucagon to work correctly in diabetes. This leads to high blood sugars right after a meal.

It is very difficult to have normal blood sugars when someone has diabetes. This may be due to another hormone called amylin. This hormone may be too low in people with Type 1 diabetes. Amylin is made in the pancreas (the part of the body that makes insulin). Amylin works by lowering blood sugars after a meal. Pramlintide is the name of the study drug. It is the man-made form of amylin. It is given as a shot (under the skin) like insulin. Pramlintide has been FDA approved.

Studies in adults have shown that amylin lowers the high levels of glucagon made after a meal. This results in improved "after meal" high blood sugars and overall blood sugar control. Currently, the drug is given as a separate shot from insulin. When given as a shot (one dose shot given all at once) to children and young adults, it seems to cause low blood sugars right after a meal. The "slowing down" of food digestion may be the cause of the low blood sugars with pramlintide use. Another possible cause of the low blood sugars may be the way drug is being given (instant shot versus a slow infusion through a pump).

ELIGIBILITY:
Inclusion Criteria:

These children will be subjects of the Texas Children's Hospital Diabetes Care Center. The subjects must be

1. 13-22 years of age at the time of enrollment.
2. Have been diagnosed with diabetes for at least 1 year and in good control (HbA1C less than or equal to 8.5%).
3. Be on continuous subcutaneous insulin infusion using an insulin pump.
4. Subjects must be otherwise healthy except for their T1DM and treated hypothyroidism.
5. Menstruating women must have a negative pregnancy test.
6. Hemoglobin equal to or greater than 12 g/dL before each study.
7. Weight more than 44 kg. -

Exclusion Criteria:

1. Age greater than 23 years or less than 13 years at the time of study
2. Any chronic disease: leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, etc or on treatment that might directly or indirectly affect glucose homeostasis, except for diabetes and hypothyroidism stable on medications
3. Anemia (hemoglobin less than 12mg/dl)
4. Lack of a supportive family environment
5. Positive pregnancy test in menstruating young women
6. Evidence or history of chemical abuse
7. Hgb A1C greater than 8.5 % in a diabetic subject
8. BMI > 90 % tile for age or < 10 % tile for age
9. Weight less than 44 kg. -

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve for glucose | 4 hrs

SECONDARY OUTCOMES:
glucagon and gastric emptying | 4 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Heptulla RA, Rodriguez LM, Bomgaars L, Haymond MW. The role of amylin and glucagon in the dampening of glycemic excursions in children with type 1 diabetes. Diabetes. 2005 Apr;54(4):1100-7. doi: 10.2337/diabetes.54.4.1100. PMID 15793249
- [Derived] Heptulla RA, Rodriguez LM, Mason KJ, Haymond MW. Twenty-four-hour simultaneous subcutaneous Basal-bolus administration of insulin and amylin in adolescents with type 1 diabetes decreases postprandial hyperglycemia. J Clin Endocrinol Metab. 2009 May;94(5):1608-11. doi: 10.1210/jc.2008-2580. Epub 2009 Feb 3. PMID 19190104